CLINICAL TRIAL: NCT00821093
Title: A 12 Week Treatment, Multi-center, Randomized, Parallel Group, Double Blind, Double Dummy Study to Assess the Superiority of Indacaterol (150 µg o.d.) Via a SDDPI in Patients With Moderate to Severe COPD, Using Salmeterol (50 µg b.i.d.) as an Active Comparator Delivered Via a DISKUS Inhaler
Brief Title: Safety and Efficacy of Indacaterol Once Daily Versus Salmeterol Twice Daily in Chronic Obstructive Pulmonary Disease (COPD)
Acronym: INSIST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CQAB149B2349; 2008-005146-23 (EudraCT Number)
Record Dates: First submitted 2009-01-09; First posted 2009-01-13 (Estimated); Results first posted 2011-08-18 (Estimated); Last update posted 2011-08-18 (Estimated); Status verified 2011-07

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: respiratory; dyspnea; breathlessness; COPD; indacaterol; long-acting β2-agonist
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea | interventions — indacaterol; Salmeterol Xinafoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Indacaterol 150 µg (Experimental): Patients inhaled indacaterol 150 μg once daily in the morning between 8:00 and 11:00 AM via a single-dose dry-powder inhaler (SDDPI) for 12 weeks. Patients also inhaled placebo to salmeterol twice daily, once in the morning between 8:00 and 11:00 AM and once in the evening between 8:00 and 11:00 PM via the manufacturer's proprietary multi-dose dry-powder inhaler (MDDPI, [DISKUS]) for 12 weeks. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol 150 µg; Drug: Placebo to salmeterol
- Salmeterol 50 µg (Active Comparator): Patients inhaled salmeterol 50 μg twice daily, once in the morning between 8:00 and 11:00 AM and once in the evening between 8:00 and 11:00 PM via the manufacturer's proprietary multi-dose dry-powder inhaler (MDDPI, [DISKUS]) for 12 weeks. Patients also inhaled placebo to indacaterol once daily in the morning between 8:00 and 11:00 AM via a single-dose dry-powder inhaler (SDDPI) for 12 weeks. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
  Interventions: Drug: Salmeterol 50 µg; Drug: Placebo to indacaterol

INTERVENTIONS:
Drug: Indacaterol 150 µg — Indacaterol 150 μg was provided in powder-filled capsules with a single-dose dry-powder inhaler (SDDPI).
  Arms: Indacaterol 150 µg
Drug: Salmeterol 50 µg — Salmeterol 50 μg was provided in the manufacturer's proprietary multi-dose dry-powder inhaler (MDDPI, [DISKUS]).
  Arms: Salmeterol 50 µg
Drug: Placebo to indacaterol — Placebo to indacaterol was provided in powder-filled capsules with a single-dose dry-powder inhaler (SDDPI).
  Arms: Salmeterol 50 µg
Drug: Placebo to salmeterol — Placebo to salmeterol was provided in the manufacturer's proprietary multi-dose dry-powder inhaler (MDDPI, [DISKUS]).
  Arms: Indacaterol 150 µg

SUMMARY:
This study compared the safety and efficacy of indacaterol 150 µg taken once daily (o.d.) versus salmeterol 50 µg taken twice daily (b.i.d) in patients 40 years old or older with chronic obstructive pulmonary disease.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥ 40 years
* Diagnosis of chronic obstructive pulmonary disease (COPD) (moderate to severe as classified by the GOLD Guidelines, 2007) and:

  * Smoking history of at least 10 pack years
  * Post-bronchodilator forced expiratory volume in 1 second (FEV1) < 80% and ≥ 30% of the predicted normal value at screening
  * Post-bronchodilator FEV1/FVC (forced vital capacity) < 70% at screening

Exclusion Criteria:

* Patients who have received systemic corticosteroids for a COPD exacerbation in the 6 weeks prior to screening or during the run-in period
* Patients requiring long-term oxygen therapy (> 15 h a day) for chronic hypoxemia
* Patients who have had a respiratory tract infection within 6 weeks prior to screening
* Patients with concomitant pulmonary disease
* Patients with a history of asthma
* Patients with diabetes Type I or uncontrolled diabetes Type II
* Any patient with lung cancer or a history of lung cancer
* Any patient with active cancer or a history of cancer with less than 5 years disease-free survival time
* Patients with a history of long QT syndrome or whose QTc interval (Fridericia's) measured at screening is prolonged
* Patients who have been vaccinated with live attenuated vaccines within 30 days prior to screening or during the run-in period
* Patients unable to successfully use a dry powder inhaler device or perform spirometry measurements

Other protocol-defined inclusion/exclusion criteria applied to the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1123 (Actual)
Dates: Start 2009-01; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceticals, Study Director — Novartis Pharmaceuticals
Locations (142):
- United States (72):
  - Novartis Investigator Site, Anniston, Alabama
  - Novartis Investigator Site, Fairhope, Alabama
  - Novartis Investigator Site, Jasper, Alabama
  - Novartis Investigator Site, Mobile, Alabama
  - Novartis Investigator Site, Glendale, Arizona
  - Novartis Investigator Site, Phoenix, Arizona
  - Novartis Investigator Site, Buena Park, California
  - Novartis Investigator Site, Encinitas, California
  - Novartis Investigator Site, Fullerton, California
  - Novartis Investigator Site, Rancho Mirage, California
  - Novartis Investigator Site, Riverside, California
  - Novartis Investigator Site, San Diego, California
  - Novartis Investigator Site, Torrance, California
  - Novartis Investigator Site, Walnut Creek, California
  - Novartis Investigator Site, Fort Collins, Colorado
  - Novartis Investigative Site, Wheat Ridge, Colorado
  - Novartis Investigative Site, Stamford, Connecticut
  - Novartis Investigative Site, Newark, Delaware
  - Novartis Investigative Center, Clearwater, Florida
  - Novartis Investigative Site, Pensacola, Florida
  - Novartis Investigative Site, South Miami, Florida
  - Novartis Investigative Site, Tamarac, Florida
  - Novartis Investigative Site, Tampa, Florida
  - Novartis Investigative Site, Marietta, Georgia
  - Novartis Investigator Site, Normal, Illinois
  - Novartis Investigator Site, River Forest, Illinois
  - Novartis Investigator Site, Skokie, Illinois
  - Novartis Investigator Site, Olathe, Kansas
  - Novartis Investigator Site, Wichita, Kansas
  - Novartis Investigator Site, Madisonville, Kentucky
  - Novartis Investigator Site, New Orleans, Louisiana
  - Novartis Investigator Site, Opelousas, Louisiana
  - Novartis Investigative Site, Baltimore, Maryland
  - Novartis Investigator Site, Ann Arbor, Michigan
  - Novartis Investigator Site, Livonia, Michigan
  - Novartis Investigator Site, Minneapolis, Minnesota
  - Novartis Investigator Site, Saint Charles, Missouri
  - Novartis Investigator Site, St Louis, Missouri
  - Novartis Investigator Site, Lincoln, Nebraska
  - Novartis Investigator Site, Omaha, Nebraska
  - Novartis Investigator Site, Henderson, Nevada
  - Novartis Investigative Site, Reno, Nevada
  - Novartis Investigative Site, Cherry Hill, New Jersey
  - Novartis Investigative Site, Summit, New Jersey
  - Novartis Investigator Site, Albuquerque, New Mexico
  - Novartis Investigative Site, Larchmont, New York
  - Novartis Investigative Site, Charlotte, North Carolina
  - Novartis Investigative Site, Hickory, North Carolina
  - Novartis Investigative Site, Raleigh, North Carolina
  - Novartis Investigative Site, Shelby, North Carolina
  - Novartis Investigator Site, Cincinnati, Ohio
  - Novartis Investigator Site, Columbus, Ohio
  - Novartis Investigator Site, Willoughby Hills, Ohio
  - Novartis Investigator Site, Tulsa, Oklahoma
  - Novartis Investigator Site, Eugene, Oregon
  - Novartis Investigator Site, Medford, Oregon
  - Novartis Investigator Site, Portland, Oregon
  - Novartis Investigative Site, Erie, Pennsylvania
  - Novartis Investigative Site, Charleston, South Carolina
  - Novartis Investigative Site, Greenville, South Carolina
  - Novartis Investigative Site, North Charleston, South Carolina
  - Novartis Investigative site, Spartanburg, South Carolina
  - Novartis Investigative Site, Union, South Carolina
  - Novartis Investigator Site, El Paso, Texas
  - Novartis Investigator Site, Fort Worth, Texas
  - Novartis Investigator Site, Houston, Texas
  - Novartis Investigator Site, San Antonio, Texas
  - Novartis Investigative Site, Abingdon, Virginia
  - Novartis Investigative Site, Richmond, Virginia
  - Novartis Investigator Site, Spokane, Washington
  - Novartis Investigator Site, Tacoma, Washington
  - Novartis Investigator Site, Milwaukee, Wisconsin
- Czechia (8):
  - Novartis Investigator Site, Cvikov
  - Novartis Investigator Site, Kyjov
  - Novartis Investigator Site, Lovosice
  - Novartis Investigator Site, Neratovice
  - Novartis Investigator Site, Ostrava
  - Novartis Investigator Site, Pardubice
  - Novartis Investigator Site, Prague
  - Novartis Investigator Site, Teplice
- Germany (25):
  - Novartis Investigative Site, Aschaffenburg
  - Novartis Investigative Site, Augsburg
  - Novartis Investigative Site, Backnang
  - Novartis Investigative Site, Berlin
  - Novartis Investigator Site, Berlin
  - Novartis Investigative Site, Bielefeld
  - Novartis Investigative Site, Borstel
  - Novartis Investigative Site, Dortmund
  - Novartis Investigative Site, Duisburg
  - Novartis Investigator Site, Frankfurt
  - Novartis Investigative Site, Geesthacht
  - Novartis Investigative Site, Hagen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Karlsruhe
  - Novartis Investigative Site, Kiel
  - Novartis Investigator Site, Leipzig
  - Novartis Investigative Site, Lübeck
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Marburg
  - Novartis Investigative Site, Neumünster
  - Novartis Investigative SIte, Oschersleben
  - Novartis Investigative Site, Rüdersdorf
  - Novartis Investigative Site, Weyhe
  - Novartis Investigative Site, Wiesloch
  - Novartis Investgative Site, Witten
- Hungary (7):
  - Novartis Investigator Site, Budapest
  - Novartis Investigator Site, Debrecen
  - Novartis Investigative Site, Deszk
  - Novartis Investigator Site, Mosonmagyaróvár
  - Novartis Investigator Site, Nyíregyháza
  - Novartis Investigator Site, Tatabánya
  - Novartis Investigator Site, Törökbálint
- India (8):
  - Novartis Investigator Site, Chennai
  - Novartis Investigator Site, Hyderabad
  - Novartis Investigator Site, Jaipur
  - Novartis Investigator Site, Mangalore
  - Novartis Investigator Site, Panjim
  - Novartis Investigator Site, Pune
  - Novartis Investigator Site, Trivandrum
  - Novartis Investigator Site, Vellore
- Slovakia (7):
  - Novartis Investigative Site, Bojnice
  - Novartis Investigator Site, Bratislava
  - Novartis Investigative Site, Humenné
  - Novartis Investigative Site, Košice
  - Novartis Investigator Site, Liptovský Hrádok
  - Novartis Investigative Site, Partizánske
  - Novartis Investigative Site, Spišská Nová Ves
- Spain (8):
  - Novartis Investigative Site, A Coruña
  - Novartis Investigator Site, Alicante
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Cáceres
  - Novartis Investigative Site, Córdoba
  - Novartis Investigative Site, Mérida
  - Novartis Investigative Site, Ourense
  - Novartis Investigative Site, Valencia
- Turkey (Türkiye) (7):
  - Novartis Investigative Site, Altunizade
  - Novartis Investigator Site, Istanbul
  - Novartis Investigator Site, Izmir
  - Novartis Investigator Site, Kartal/Istanbul
  - Novartis Investigative Site, Kinikli / Denizli
  - Novartis Investigative Site, Mersin
  - Novartis Investigator Site, Yenisehir/Izmir

REFERENCES:
- [Derived] Korn S, Kerwin E, Atis S, Amos C, Owen R, Lassen C; INSIST study group. Indacaterol once-daily provides superior efficacy to salmeterol twice-daily in COPD: a 12-week study. Respir Med. 2011 May;105(5):719-26. doi: 10.1016/j.rmed.2011.02.008. Epub 2011 Mar 1. PMID 21367594

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of total 1123 randomized patients, two patients withdrew from study prior to exposure to study drug.
Groups:
- Indacaterol 150 μg: Patients inhaled indacaterol 150 μg once daily in the morning between 8:00 and 11:00 AM via a single-dose dry-powder inhaler (SDDPI) for 12 weeks. Patients also inhaled placebo to salmeterol twice daily, once in the morning between 8:00 and 11:00 AM and once in the evening between 8:00 and 11:00 PM via the manufacturer's proprietary multi-dose dry-powder inhaler (MDDPI, [DISKUS]) for 12 weeks. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
- Salmeterol 50 μg: Patients inhaled salmeterol 50 μg twice daily, once in the morning between 8:00 and 11:00 AM and once in the evening between 8:00 and 11:00 PM via the manufacturer's proprietary multi-dose dry-powder inhaler (MDDPI, [DISKUS]) for 12 weeks. Patients also inhaled placebo to indacaterol once daily in the morning between 8:00 and 11:00 AM via a single-dose dry-powder inhaler (SDDPI) for 12 weeks. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
Period: Overall Study
Arm/Group | Indacaterol 150 μg | Salmeterol 50 μg
Started | 560 | 563
Exposed to Drug | 559 | 562
Completed | 511 | 523
Not Completed | 49 | 40
Not completed — Adverse Event | 20 | 12
Not completed — Withdrawal by Subject | 9 | 13
Not completed — Lost to Follow-up | 9 | 3
Not completed — Protocol deviation | 3 | 6
Not completed — Abnormal laboratory value(s) | 2 | 0
Not completed — Lack of Efficacy | 2 | 2
Not completed — Death | 2 | 1
Not completed — Abnormal test procedure result(s) | 1 | 1
Not completed — Administrative problems | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Indacaterol 150 μg | Salmeterol 50 μg | Total
Number analyzed (Participants) | 559 | 562 | 1121
Age Continuous [Mean (Standard Deviation); unit: years] — Demographic data are based on the safety set of patients.
  years | 62.4 (8.86) | 63.2 (8.69) | 62.8 (8.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 189 | 147 | 336
  Male | 370 | 415 | 785

OUTCOME MEASURES:

1. Primary Outcome: Forced Expiratory Volume in 1 Second (FEV1) Standardized (With Respect to Time) Area Under the Curve (AUC) From 5 Minutes to 11 Hours 45 Minutes Post-dose at the End of the Study (Week 12, Day 84)
Description: FEV1 was measured with spirometry conducted according to internationally accepted standards. Measurements were made at 5 and 30 minutes; 1, 2, 3, 4, and 8 hours; 11 hours 10 minutes and 11 hours 45 minutes post-dose at the end of the study (Week 12, Day 84). Standardized FEV1 AUC was calculated by the trapezoidal rule. The analysis included baseline FEV1 and FEV1 pre-dose and 10-15 minutes post-dose of salbutamol/albuterol during screening as covariates.
Time Frame: From 5 minutes to 11 hours 45 minutes post-dose at the end of the study (Week 12, Day 84)
Population: Full analysis set: All randomized patients who received at least 1 dose of study drug, last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol 150 μg | Salmeterol 50 μg
Number analyzed (Participants) | 504 | 488
Liters | 1.47 (0.009) | 1.41 (0.010)

2. Secondary Outcome: Trough Forced Expiratory Volume in 1 Second (FEV1) 24 Hours Post-dose at the End of the Study (Week 12 + 1 Day, Day 85)
Description: FEV1 was measured with spirometry conducted according to internationally accepted standards. Trough FEV1 was defined as the average of measurements made 23 hours 10 minutes and 23 hours 45 minutes post-dose at the end of treatment. The analysis included baseline FEV1 and FEV1 pre-dose and 10-15 minutes post-dose of salbutamol/albuterol during screening as covariates.
Time Frame: 24 hours post-dose at the end of the study (Week 12 + 1 day, Day 85)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol 150 μg | Salmeterol 50 μg
Number analyzed (Participants) | 522 | 512
Liters | 1.41 (0.009) | 1.35 (0.010)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: The Safety set included all patients who received at least one dose of study drug.
Arm/Group | Indacaterol 150 μg | Salmeterol 50 μg
Serious Adverse Events (participants affected / at risk) | 20/559 | 16/562
Other Adverse Events (participants affected / at risk) | 0/559 | 0/562
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol 150 μg (N=559) | Salmeterol 50 μg (N=562)
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 2 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Contrast media allergy (Immune system disorders) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Upper respiratory tract infection bacterial (Infections and infestations) | 2 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0
Weight decreased (Investigations) | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Hemiparesis (Nervous system disorders) | 1 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0
Radicular syndrome (Nervous system disorders) | 0 | 1
Spinal cord compression (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4 | 7
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.